CLINICAL TRIAL: NCT00402532
Title: Immunosuppressive Therapy With Certican (Everolimus) After Lung Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Martin Strueber, Martin Strueber, MD, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ever-Lung-DE01/RAD-LungDE01
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Immunosuppression; Mortality; Graft rejection; Bronchiolitis obliterans; Opportunistic infections; Nephrotoxicity
MeSH Terms: conditions — Bronchiolitis Obliterans; Opportunistic Infections | interventions — Everolimus; Mycophenolic Acid

ARMS (2):
- Everolimus (Active Comparator)
  Interventions: Drug: Everolimus
- Mycophenolatmofetil (Active Comparator)
  Interventions: Drug: Mycophenolatmofetil

INTERVENTIONS:
Drug: Everolimus — Initial dosage 2 x 0.75 mg/d
  Other Names: Certican
  Arms: Everolimus
Drug: Mycophenolatmofetil — Initial dosage 2 x 500 mg/d intravenous
  Other Names: Cellcept
  Arms: Mycophenolatmofetil

SUMMARY:
The purpose of this study is to determine whether Everolimus is effective in the treatment and prevention of chronic graft dysfunction and chronic graft rejection after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of Single or Bilateral Lung Transplantation
* Informed consent
* Recipients who are able to receive Everolimus at week 3 after Lung Transplantation
* women of childbearing potential must have a negative pregnancy test within 48 hours of enrolment
* women of childbearing potential must use appropriate contraceptive method at enrolment, during the study and up to 8 weeks after the end of the study
* donor must not have relevant pulmonary diseases
* donor must have oxygen partial pressure higher than 300 mmHg at FiO 1.0 and positive end-expiratory pressure of 5 cm H2O.

Exclusion Criteria:

* systemic infection of the donor
* donor: signs or symptoms of aspiration
* donor: severe pulmonary injury or contusion
* donor: malignant neoplasm of the lung
* donor: HIV positive
* recipients who receive immunosuppressive agents not used in this protocol
* recipients who participated within 30 days before study start or are currently participating in another investigational drug trial
* HIV positive recipient
* systemic infection of the recipient
* recipients of combined/ multiple transplantations
* pregnancy of the recipient
* recipients with signs/ Symptoms of impaired wound healing of the pulmonary anastomoses
* recipients who are still on artificial respiration or who are not able to swallow tablets at week 3 after transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2005-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of bronchiolitis obliterans syndrome and mortality and need for change of immunosuppressive medication within 2 years from transplantation | 2 years

SECONDARY OUTCOMES:
Incidence and severity of Nephrotoxicity within 2 years of transplantation | 2 years
Incidence and severity of opportunistic infections within 2 years of transplantation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Strueber, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Division of Thoracic and Cardiovascular Surgery, Hanover, Germany